CLINICAL TRIAL: NCT00892866
Title: Comparative Analysis of CA-IX, p16, Proliferative Markers, and Human Papilloma Virus (HPV) in the Diagnosis of Significant Cervical Lesions in Patients With a Cytologic Diagnosis of Atypical Glandular Cells (AGC)
Brief Title: CA-IX, p16, Proliferative Markers, and HPV in Diagnosing Cervical Lesions in Patients With Abnormal Cervical Cells
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GOG Foundation (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: GOG-0237; NCI-2009-01103 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000632236; GOG-0237 (Other: Gynecologic Oncology Group); GOG-0237 (Other: DCP); GOG-0237 (Other: CTEP); N01CM62201 (NIH); U10CA101165 (NIH); UG1CA189867 (NIH)
Record Dates: First submitted 2009-05-02; First posted 2009-05-05 (Estimated); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Atypical Endometrial Hyperplasia; Human Papillomavirus Infection; Stage 0 Cervical Cancer AJCC v7
MeSH Terms: conditions — Endometrial Hyperplasia; Papillomavirus Infections; Uterine Cervical Dysplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ancillary-Correlative (biomarkers in cervical cancer) (Other): Patients undergo liquid-based cytology specimen sample collection for analysis of CA-IX, p16, Ki-67, and MCM2 expression via IHC and for the presence of high risk HPV DNA and HPV genotyping.
  Interventions: Other: Cytology Specimen Collection Procedure; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Other: Cytology Specimen Collection Procedure — Correlative studies
  Other Names: Cytologic Sampling
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This research trial studies carbonic anhydrase 9 (CA-IX), p16, proliferative markers, and human papilloma virus (HPV) in diagnosing cervical lesions in patients with abnormal cervical cells. Studying biomarkers in abnormal cervical cells may improve the ability to find cervical lesions and plan effective treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To examine CA-IX, p16, Ki-67, and mini-chromosome maintenance complex component 2 (MCM2) expression in liquid-based cytology (LBC) specimens to see which subset of markers can provide the optimal diagnosis of significant cervical lesions in women in North America with a cytologic diagnosis of atypical glandular cells (AGC) and a positive test for high risk human papillomavirus (HPV).

II. To examine high risk HPV, CA-IX, p16, Ki-67, and MCM2 expression in LBC specimens to see which subset of markers can provide the optimal diagnosis of significant cervical lesions in women in Japan and Korea (with each country's cohort analyzed separately) with a cytologic diagnosis of AGC.

SECONDARY OBJECTIVES:

I. To determine whether the accuracy of diagnosis based on high risk HPV and expression of CA-IX, p16, Ki-67, and/or MCM2 varies with patient age at enrollment and country of enrollment.

TERTIARY OBJECTIVES:

I. To assess biomarker expression, loss of heterozygosity, and chromosome gains/losses in formalin-fixed, paraffin-embedded tissue from the highest grade or most abnormal lesion in women from North America, Japan, or Korea presenting with a cytologic diagnosis of AGC or with a cytologic/histologic diagnosis of adenocarcinoma in situ (AIS).

II. To determine CA-IX, p16, Ki67, and MCM2 expression in LBC specimens to see which subset (or combination) of markers will provide higher sensitivity in the diagnosis of cervical adenocarcinoma in situ (AIS).

OUTLINE:

Patients undergo liquid-based cytology specimen sample collection for analysis of CA-IX, p16, Ki-67, and MCM2 expression via immunohistochemistry (IHC) and for the presence of high risk HPV deoxyribonucleic acid (DNA) and HPV genotyping.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a cytologic diagnosis of AGC (AGC, atypical endocervical cells [AEC], atypical endometrial cells [AEmC]) or a cytologic/histologic diagnosis of AIS documented within the last 6 months who can wait at least one week after the AGC or AIS diagnosis to have an LBC specimen (i.e., ThinPrep) collected and then receive any other intervention; acceptable time frame range is 4 days prior to registration to 7 days after registration
* Patients with positive HPV results who are willing to undergo a complete histologic examination of the uterus and cervix, including the cervical transformation zone, within 6 months of the AGC or AIS diagnosis (histologic examination includes a loop electrosurgical excision procedure [LEEP], loop excision of the transformation zone [LETZ], excisional cone biopsy, or hysterectomy)
* Patients must have signed an approved informed consent and authorization permitting release of personal health information

Exclusion Criteria:

* Patients who have had a hysterectomy
* History of endometrial hyperplasia or cancer of the endometrium, vagina, or cervix
* Patients who have previously been treated, or are currently being treated with radiation therapy or chemotherapy for vaginal or cervical cancer
* Patients who are known to be human immunodeficiency virus (HIV)-positive
* Patients who are pregnant and thought to be at risk for excessive bleeding or preterm labor if a cone biopsy is performed

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 877 (Estimated)
Dates: Start 2009-04-13 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Biomarker expression in patients from North America | Baseline
  CA-IX, p16, Ki-67, and MCM2 expression in LBC specimens is measured via IHC. A logistic regression and receiver operating characteristic (ROC)-type analysis will be performed.
Biomarker expression in patients from Japan | Baseline
  CA-IX, p16, Ki-67, and MCM2 expression in LBC specimens is measured via IHC. A logistic regression and ROC-type analysis will be performed.
Biomarker expression in patients from Korea | Baseline
  CA-IX, p16, Ki-67, and MCM2 expression in LBC specimens is measured via IHC. A logistic regression and ROC-type analysis will be performed.

SECONDARY OUTCOMES:
Effect of patient age on the accuracy of diagnosis based on CA-IX, HPV, p16, Ki-67, and/or MCM2 expression in the North American population | Baseline
  Logistic regression analyses will be performed to assess the effect of age and country on sensitivity, specificity, false positive rate (FPR), and complement negative predictive value (NPVC.). For each country and at each age, an upper 95% confidence limit will be calculated for the NPVC.
Effect of patient age on the accuracy of diagnosis based on CA-IX, HPV, p16, Ki-67, and/or MCM2 expression in the Korean and Japanese populations | Baseline
  Logistic regression analyses will be performed to assess the effect of age and country on sensitivity, specificity, FPR, and NPVC. For each country and at each age, an upper 95% confidence limit will be calculated for the NPVC.

OTHER OUTCOMES:
Biomarker expression, loss of heterozygosity (LOH), chromosome gains, and chromosome losses in tissue from the highest grade or most abnormal lesions in women with AGC | Baseline
  Exploratory analyses of genomic alterations, including LOH as well as chromosome gains and chromosome losses will be performed to identify genomic alterations associated with cervical dysplasia/neoplasia.
CA-IX expression, combined p16 and Ki67 expression, and MCM2 expression in LBC specimens | Baseline
  Will be used to see which subset of markers will provide the higher and sensitivity in the diagnosis of cervical AIS.

CONTACTS AND LOCATIONS:
Overall Officials: Shu-Yuan liao, Principal Investigator — Gynecologic Oncology Group
Locations (163):
- United States (135):
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California
  - Saint Joseph Hospital - Orange, Orange, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Olive View-University of California Los Angeles Medical Center, Sylmar, California
  - Hartford Hospital, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Alphonsus Medical Center-Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Cancer Clinic, Sandpoint, Idaho
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Elkhart Clinic, Elkhart, Indiana
  - Michiana Hematology Oncology PC-Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - IU Health La Porte Hospital, La Porte, Indiana
  - Michiana Hematology Oncology PC-Mishawaka, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - Michiana Hematology Oncology PC-Plymouth, Plymouth, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology Oncology PC-South Bend, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - Michiana Hematology Oncology PC-Westville, Westville, Indiana
  - Providence Medical Center, Kansas City, Kansas
  - Kansas Institute of Medicine Cancer and Blood Center, Lenexa, Kansas
  - Minimally Invasive Surgery Hospital, Lenexa, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Advent Health - Shawnee Mission Medical Center, Shawnee Mission, Kansas
  - Woman's Hospital, Baton Rouge, Louisiana
  - Maine Medical Center-Bramhall Campus, Portland, Maine
  - Maine Medical Center- Scarborough Campus, Scarborough, Maine
  - Baystate Medical Center, Springfield, Massachusetts
  - Lakeland Hospital Niles, Niles, Michigan
  - William Beaumont Hospital-Royal Oak, Royal Oak, Michigan
  - Lakeland Medical Center Saint Joseph, Saint Joseph, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Centerpoint Medical Center LLC, Independence, Missouri
  - Truman Medical Centers, Kansas City, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Saint Joseph Health Center, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Heartland Hematology and Oncology Associates Incorporated, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Radiation Oncology Center, Liberty, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Saint Joseph Oncology Inc, Saint Joseph, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Hospital, Missoula, Montana
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Women's Cancer Center of Nevada, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Norris Cotton Cancer Center-Nashua, Nashua, New Hampshire
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - FirstHealth of the Carolinas-Moore Regional Hospital, Pinehurst, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Delaware Radiation Oncology, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Dublin Methodist Hospital, Dublin, Ohio
  - Central Ohio Breast and Endocrine Surgery, Gahanna, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - OhioHealth Mansfield Hospital, Mansfield, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - OhioHealth Marion General Hospital, Marion, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Saint Alphonsus Medical Center-Baker City, Baker City, Oregon
  - Saint Alphonsus Medical Center-Ontario, Ontario, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Geisinger Cancer Services-Pottsville, Pottsville, Pennsylvania
  - Community Medical Center, Scranton, Pennsylvania
  - Geisinger Medical Oncology-Selinsgrove, Selinsgrove, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - University of Texas Medical Branch, Galveston, Texas
  - Memorial Hermann Texas Medical Center, Houston, Texas
  - UTMB Cancer Center at Victory Lakes, League City, Texas
  - Big Horn Basin Cancer Center, Cody, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming
- Japan (17):
  - Tohoku University School of Medicine, Sendai, Aoba-ku
  - Kure National Hospital, Kure, Hiroshima
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Hyogo Cancer Center, Akashi, Hyōgo
  - Iwate Medical University Hospital, Shiwa-gun, Iwate
  - Kagoshima City Hospital, Kagoshima, Kagoshima-ken
  - Niigata University Medical and Dental Hospital, Niigata, Niigata
  - University of the Ryukyus Hospital-Col Health Scnc, Nakagami-gun, Okinawa
  - Keio University, Shinjuku-ku, Tokyo
  - Hiroshima University Hospital, Hiroshima
  - Shikoku Cancer Center, Matsuyama
  - National Kyushu Cancer Center, Minamiku
  - Jikei University School of Medicine, Minato-ku, Tokyo
  - Kindai University, Osaka
  - Saitama Medical University International Medical Center, Saitama
  - National Cancer Center Hospital, Tokyo
  - Tottori University, Tottori
- South Korea (11):
  - Keimyung University-Dongsan Medical Center, Dalseo-gu, Daegu
  - National Cancer Center-Korea, Goyang-si, Gyeonggi-do
  - Inha University, Jung-gu, Incheon
  - Catholic University of Korea-Seoul Saint Mary's Hospital, Seoul, Korea
  - Seoul National University Bundang Hospital, Seongnam, Kyeonggi-do
  - Gachon University Gil Hospital, Incheon
  - Asan Medical Center, Seoul
  - Gangnam Severance Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Yonsei University Health System-Severance Hospital, Seoul
  - Kyung Hee University Hospital at Gangdong, Seoul